CLINICAL TRIAL: NCT03757169
Title: Effect of Isometric Hand Grip Training on Blood Pressure of Hypertensive Patients With Obstructive Sleep Apnea
Brief Title: Isometric Hand Grip Training in Obstructive Sleep Apnea (OSA)
Acronym: OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pinto Pedrosa, Head of sleep laboratory and heart emergency room of Pernambuco , Principal Investigator., University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: isopress03
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: training; hand grip; exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: There are two randomized groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Verbal informations about the disease, and exercise behavior, and nutrition.
  Interventions: Other: Control
- Hand grip group (Active Comparator): Three supervised sessions por week: 4 series (2 at each arm) of two minutes of isometric hand grip contraction at 30% of maximal voluntary contraction. Between series there will be two minutes to rest.
  Interventions: Other: Hand grip isometric contraction

INTERVENTIONS:
Other: Hand grip isometric contraction — The patients at the Hand Grip group will perform 12 weeks of hand grip exercises, three times/week for 16 minutes with time to rest.
  Arms: Hand grip group
Other: Control — The patients will receive verbal orientations about the OSA and the arterial hypertension.
  Arms: Control group

SUMMARY:
Obstructive sleep apnea (OSA) is a common clinical condition, involving the development of arterial hypertension. A Meta analysis study have shown that isometric hand grip training promotes blood pressure reduction. It is going to be conducted a clinical trail to determine the effects of hand grip training in OSA patients to change the arterial hypertension.

DETAILED DESCRIPTION:
Background: obstructive sleep apnea (OSA) is a common clinical condition, involving the development of arterial hypertension. Meta analysis study have shown that isometric hand grip strength promotes blood pressure reduction, and its reduction is higher than that observed after aerobic training. Objective: to analyze the effects of the isometric hand grip on blood pressure changes of patients with uncontrolled arterial hypertension with OSA. Methods: a randomized controlled trial involving 18 adults with OSA and uncontrolled arterial hypertension of both sexes, randomized between control group (receive general guidelines) and hand grip group. 12 weeks of training with load equivalent to 30% of maximum voluntary capacity was performed. All participants will be submitted for evaluation of blood pressure (BP) central and brachial, pulse wave velocity, full polysomnography,before and after the study protocol (the change from the baseline at 12 weeks). Expected results: the authors believe that hand grip training can change (reduce) blood pressure in patient with OSA.

ELIGIBILITY:
Inclusion Criteria:

* OSA diagnose based on polysomnography,
* Apnea-Hypopnea Index (AHI) > 5,
* arterial hypertension (systolic arterial pressure > 140 mmHg or diastolic arterial pressure > 90 mmHg)

Exclusion Criteria:

* other heart disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change at ambulatory blood pressure monitoring | Change from the baseline ambulatory blood pressure monitoring at 12 weeks
  24h of monitoring blood pressure

SECONDARY OUTCOMES:
Change at blood pressure | Change from the baseline brachial blood pressure at 12 weeks
  Three measurement of brachial blood pressure
Chance at Apnea-Hypopnea Index (AHI) | Change from the baseline AHI at 12 weeks
  Index obtained by the Polysomnography to detect the level of Apnea-Hypopnea Index. The higher level, the worse the disease. The value of the AHI between 5 to 15 events/hour means mild disease. AHI between 16 to 30 events/hour means moderate disease, and more than 30 events/hour means severe disease.
Change at Pulse wave velocity | Change from the baseline pulse wave velocity at 12 weeks
  To evaluate the pulse wave velocity (femoral, carotid and aortic) to detect the occurrence of arterial disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Pronto Socorro Cardiológico de Pernambuco - Procape, Recife, Pernambuco, Brazil